CLINICAL TRIAL: NCT04267432
Title: The Assessment of TCI633 Probiotics on Pain Relief and Functional Improvement in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 201703132MSC
Record Dates: First submitted 2020-01-06; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- TCI633 (Experimental): Testing product
  Interventions: Dietary Supplement: TCI633
- Type 2 collagen (Active Comparator): Known drug for OA
  Interventions: Drug: Type 2 collagen

INTERVENTIONS:
Dietary Supplement: Placebo — Blank
  Arms: Placebo
Dietary Supplement: TCI633 — Probiotics
  Arms: TCI633
Drug: Type 2 collagen — Positive control group
  Arms: Type 2 collagen

SUMMARY:
To assess TCI633 probiotics on pain relief and functional improvement in osteoarthritis

DETAILED DESCRIPTION:
This is a double-blind and randomized study. Subjects are informed to consume the samples before meals in the morning every day. The clinical and radiological diagnosis of osteoarthritis of the knee is evaluated by the doctor. The blood samples and questionnaires are collected at every visit of the trial.

ELIGIBILITY:
Inclusion criteria

1. Osteoarthritis patients with joint pain or discomfort (diagnosed by the physician for severe classification of the Kellgren-Lawrence Grade 1-3)
2. Without heart, liver, kidney, endocrine and other major organic diseases (patient return)

Exclusion criteria

1. With heart, liver (GOT and GPT values are 3-fold higher than the standard maximum), kidney (estimated creatinine clearance less than 25 mL/min), endocrine and other major organic diseases (patient return)
2. People with mental illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
KL Grade (evaluated by doctor) | Change from baseline at 6 months
  Pain relief and functional improvement in osteoarthritis
WOMAC™ Osteoarthritis Index | Change from baseline at 6 months
  The questionnaire includes three-part: i) join pain (five questions); ii) joint stiffness (two questions); and, iii) physical functions of joints (seventeen questions). Each question is scored 0-4. Low to high WOMAC scores represent slight to severe OA symptoms. The lower scores mean a better outcome.

SECONDARY OUTCOMES:
Blood C-terminal telopeptide of collagen type II (CTX-II) level | Change from baseline at 6 months
  To measure the level of CTX-II in blood
Blood C-reactive protein (CRP) level | Change from baseline at 6 months
  To measure the level of CRP in blood

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Ming Wang, Doctor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan